CLINICAL TRIAL: NCT00496015
Title: Prophylactic Antipyretic Treatment in Children Receiving Booster Dose of Pneumococcal Vaccine GSK1024850A and DTPa-HBV-IPV/Hib Vaccine (Infanrix Hexa) and Assessment of Impact of Pneumococcal Vaccination on Nasopharyngeal Carriage
Brief Title: Prophylactic Antipyretic Treatment in Children Receiving Booster Dose of Pneumococcal Conjugate Vaccine GSK1024850A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107137
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2017-05

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus Pneumoniae Vaccines; Meningococcal disease; Carriage; Prophylactic antipyretic; Safety; Pneumococcal vaccine; Fever; Pneumococcal disease; Immunogenicity; Meningococcal vaccine; Booster vaccination
MeSH Terms: conditions — Streptococcal Infections; Meningococcal Infections; Fever; Pneumococcal Infections | interventions — diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; Acetaminophen

ARMS (5):
- Synflorix I Group (Experimental): Subjects were vaccinated with 3 primary vaccination doses of Synflorix™ vaccine with prophylactic administration of paracetamol in study 10PN-PD-DIT-010 (107017), and received in this study at 12-15 months of age a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa along with prophylactic antipyretic treatment.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A.; Biological: Infanrix hexa.; Drug: Paracetamol.
- Synflorix II Group (Experimental): Subjects were vaccinated with 3 primary vaccination doses of Synforix™ vaccine without prophylactic administration of paracetamol in study 10PN-PD-DIT-010 (107017), and received in this study at 12-15 months of age a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa without prophylactic antipyretic treatment
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A.; Biological: Infanrix hexa.
- Synflorix PRE Group (Experimental): Subjects were vaccinated with 3 primary vaccination doses of Synforix™ vaccine without prophylactic administration of paracetamol in study 10PN-PD-DIT-010 (107017), and received in this study (before the implementation of the protocol amendment) at 12-15 months of age a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa without prophylactic antipyretic treatment.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A.; Biological: Infanrix hexa.
- Synflorix POST Group (Experimental): Subjects were vaccinated with 3 primary vaccination doses of Synforix™ vaccine without prophylactic administration of paracetamol in study 10PN-PD-DIT-010 (107017), and received in this study (after the implementation of the protocol amendment) at 12-15 months of age a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa without prophylactic antipyretic treatment.
  Interventions: Biological: Pneumococcal conjugate vaccine GSK1024850A.; Biological: Infanrix hexa.
- Mencevax + Infanrix Hexa Group (Active Comparator): Age-matched pneumococcal vaccine unprimed group receiving a single dose of Mencevax™ vaccine co-administered with Infanrix™ hexa vaccine.
  Interventions: Biological: Infanrix hexa.; Biological: Meningococcal vaccine GSK134612.

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK1024850A. — 1 intramuscular injection.
  Arms: Synflorix I Group; Synflorix II Group; Synflorix POST Group; Synflorix PRE Group
Biological: Infanrix hexa. — 1 intramuscular injection.
  Other Names: DTPa-HBV-IPV/Hib
Biological: Meningococcal vaccine GSK134612. — 1 intramuscular injection.
  Other Names: Mencevax™
  Arms: Mencevax + Infanrix Hexa Group
Drug: Paracetamol. — Body weight of < 7 kg: none; Body weight of ≥ 7 kg to < 9 kg : 3 suppositories of 125 mg to be administered at 8h intervals after vaccination. Body weight of ≥ 9 kg: 4 suppositories of 125 mg to be administered at 6h intervals after vaccination.
  Arms: Synflorix I Group

SUMMARY:
The purpose of this trial is to assess if the rate of febrile reactions following the co-administration of a booster dose of pneumococcal conjugate vaccines with standard infant vaccines is lowered when paracetamol is given prophylactically and to assess the impact of pneumococcal conjugate vaccine on pneumococcal and H. influenzae nasopharyngeal carriage compared to control group receiving meningococcal conjugate vaccine (GSK134612).

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00370318).

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 12-15 months of age at the time of the vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Subjects in the unprimed group

• A male or female who previously participated in study 107017 and received 3 doses of pneumococcal conjugate vaccine GSK1024850A.

Exclusion Criteria:

For all subjects:

* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Indication, other than specified in the protocol, for prophylactic antipyretic treatment.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within one month preceding the dose of study vaccines, or planned use during the entire study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the dose of study vaccines.
* Planned administration/administration of a vaccine not foreseen by the study protocol, during the period starting one month before the dose of study vaccines and up to one month after the dose of study vaccines.
* History of, or intercurrent, diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or progressive neurological disease.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Administration of immunoglobulins and/or any blood products within three months preceding administration of the dose of study vaccines or planned administration during the study period.
* Subjects of which both parents have a history of atopia.
* Subject has received systemic antibiotic therapy for acute illness within 24 hours prior to the vaccination.
* Subject is likely to receive antipyretic treatment as a result of a concomitant illness or has been treated with paracetamol within the past 24 hours.

DTPa-HBV-IPV/Hib vaccine:

* Known hypersensitivity after previous administration of diphtheria, tetanus, pertussis, polio, hepatitis B and Hib vaccines or to any component of the vaccines.
* Encephalopathy.
* As with other vaccines, administration of DTPa-HBV-IPV/Hib should be postponed in subjects suffering from acute mild, moderate or severe illness.

For subjects in the AP-AP, AP-NAP and NAP groups:

• Administration of any pneumococcal, diphtheria, tetanus, pertussis, polio, hepatitis B and/or Haemophilus influenzae type b vaccines other than allowed and used in study 107017.

For subjects in the AP-AP group:

• Subject with any contraindication to treatment with paracetamol.

For subjects in the unprimed group:

* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W-135 and/or Y.
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroups A, C, W-135 and/or Y.
* Planned administration of a hepatitis B vaccine not foreseen by the study protocol during the period starting one month after the dose of study vaccines and up to study end.
* Previous vaccination with tetanus toxoid containing vaccines including T, DTP, DT, DTP-IPV, DTP-HBV-IPV and Hib-TT vaccines six months prior to study entry.
* History of meningococcal disease due to serogroup A, C, W, or Y.
* Administration of any pneumococcal vaccine since birth.
* Full vaccination history since birth not available.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2007-07-02 (Actual); Primary Completion 2008-03-25 (Actual); Study Completion 2009-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Czechia (8):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Znojmo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Prymula R, Siegrist CA, Chlibek R, Zemlickova H, Vackova M, Smetana J, Lommel P, Kaliskova E, Borys D, Schuerman L. Effect of prophylactic paracetamol administration at time of vaccination on febrile reactions and antibody responses in children: two open-label, randomised controlled trials. Lancet. 2009 Oct 17;374(9698):1339-50. doi: 10.1016/S0140-6736(09)61208-3. PMID 19837254
- [Background] Prymula R, Hanovcova I, Splino M, Kriz P, Motlova J, Lebedova V, Lommel P, Kaliskova E, Pascal T, Borys D, Schuerman L. Impact of the 10-valent pneumococcal non-typeable Haemophilus influenzae Protein D conjugate vaccine (PHiD-CV) on bacterial nasopharyngeal carriage. Vaccine. 2011 Feb 24;29(10):1959-67. doi: 10.1016/j.vaccine.2010.12.086. Epub 2011 Jan 6. PMID 21215830
- [Background] Prymula R et al. Does prophylactic paracetamol influence the effect of 10-valent pneumococcal non-typeable Haemophilus influenzae protein-D conjugate vaccine (PHiD-CV) on pneumococcal nasopharyngeal carriage? Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Prymula R et al. Effects on serotype 6A and 6B nasopharyngeal carriage following immunization with 10-valent pneumococcal non-typeable Haemophilus influenzae protein-D conjugate vaccine. Abstract presented at the 28th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID). Nice, France, 4-8 May 2010.
- [Background] Prymula R et al. Limited clinical benefit but reduced antibody responses to paediatric vaccines following prophylactic paracetamol administration. Abstract presented at the 4th Europaediatrics, Moscow, Russia, 03-06 July 2009.
- [Background] Prymula R et al. The 10-valent pneumococcal vaccine conjugated to protein-D (PHiD-CV) reduces nasopharyngeal carriage of Streptococcus pneumoniae (SP) vaccine serotypes in Czech children. Abstract presented at the 6th World Congress of the World Society for Pediatric Infectious Diseases (WSPID). Buenos Aires, Argentina, 19-22 November 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107137 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study with the same centers as the primary vaccination study 10PN-PD-DIT-010 (107017/NCT00370318) and all subjects enrolled in the primary vaccination study and having received Synflorix vaccine were invited to participate in the study. In addition, an age-matched pneumococcal vaccine unprimed control group has been enrolled.
Period: Overall Study
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Started | 178 | 27 | 172 | 37 | 336
Completed | 177 | 27 | 172 | 36 | 336
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Synflorix I Group: Subjects were vaccinated with 3 primary vaccination doses of Synforix™ vaccine with prophylactic administration of paracetamol in study 10PN-PD-DIT-010 (107017), and received in this study at 12-15 months of age a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa along with prophylactic antipyretic treatment.
- Total: Total of all reporting groups
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group | Total
Number analyzed (Participants) | 178 | 27 | 172 | 37 | 336 | 750
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.6 (0.77) | 13.2 (0.74) | 12.7 (0.77) | 13.1 (1.15) | 13.1 (1.1) | 12.6 (0.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 11 | 79 | 18 | 155 | 353
  Male | 88 | 16 | 93 | 19 | 181 | 397
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: White - Arabic/North African heritage | 0 | 0 | 0 | 0 | 9 | 9
  Geographic ancestry: White - Caucasian / European heritage | 177 | 27 | 172 | 37 | 327 | 740
  Geographic ancestry: Other - African + White-Caucasian | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reported With Core Fever (Rectal Temperature) Greater Than or Equal to (≥) the Cut-off
Description: The cut-off for core fever was 38.0 degrees Celsius (ºC).
Time Frame: Within 4 days (Day 0-3) after primary vaccine dose.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 178 | 27 | 172 | 37 | 336
Participants | 64 | 14 | 100 | 16 | 146
Statistical Analysis 1: Comparison: Synflorix I Group vs Synflorix PRE Group; Test type: Superiority — Superiority criteria: The lower limit (LL) of the standardized asymptotic 95% confidence interval (CI) for the difference between groups (Synflorix PRE Group minus Synflorix I Group) was above 0%; Difference in percentages = 22.18, 95% CI 2-sided [11.78 to 32.11]

2. Secondary Outcome: Number of Subjects Reported With Core Fever (Rectal Temperature) Greater Than (>) the Cut-off
Description: The cut-off value for core fever (rectal temperature) was 39.0ºC.
Time Frame: Within 4 days (Day 0-3) after primary vaccination dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 178 | 27 | 172 | 37 | 336
Participants | 4 | 0 | 14 | 1 | 16

3. Secondary Outcome: Number of Subjects Reported With Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any occurrence of the specified symptom regardless of intensity. Grade 3 pain was defined as cried when limb was moved/spontaneously painful. Grade 3 redness/swelling was defined as redness/swelling > 30 millimeters (mm) from injection site.
Time Frame: During the 4-day (Days 0-3) post-primary vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 178 | 27 | 172 | 37 | 336
Participants
  Any Pain | 54 | 10 | 79 | 19 | 114
  Grade 3 Pain | 2 | 2 | 10 | 3 | 4
  Any Redness | 89 | 9 | 74 | 12 | 146
  Grade 3 Redness | 7 | 1 | 14 | 1 | 16
  Any Swelling | 52 | 8 | 50 | 13 | 71
  Grade 3 Swelling | 2 | 1 | 9 | 3 | 12

4. Secondary Outcome: Number of Subjects Reported With Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were drowsiness, fever (rectal temperature ≥ 38.5°C), irritability and loss of appetite. Any was defined as any occurrence of the specified symptom regardless of intensity and relation to vaccination. Grade 3 drowsiness was defined as drowsiness that prevented normal activity. Grade 3 fever was defined as rectal temperature >40.0°C. Grade 3 irritability was defined as crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite was defined as not eating at all. Related was defined as solicited symptoms assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 178 | 27 | 172 | 37 | 336
Participants
  Any Drowsiness | 91 | 11 | 84 | 18 | 146
  Grade 3 Drowsiness | 0 | 0 | 1 | 1 | 2
  Related Drowsiness | 84 | 11 | 79 | 18 | 120
  Any Fever (rectal temperature ≥ 38.0°C) | 64 | 14 | 100 | 16 | 146
  Grade 3 Fever (rectal temperature > 40.0°C) | 1 | 0 | 1 | 0 | 3
  Related Fever (rectal temperature > 40.0°C) | 62 | 14 | 99 | 16 | 140
  Any Irritability | 86 | 17 | 105 | 19 | 147
  Grade 3 Irritability | 1 | 0 | 2 | 2 | 2
  Related Irritability | 80 | 17 | 98 | 18 | 129
  Any Loss of appetite | 47 | 8 | 46 | 10 | 88
  Grade 3 Loss of appetite | 0 | 0 | 4 | 1 | 3
  Related Loss of appetite | 42 | 7 | 41 | 10 | 71

5. Secondary Outcome: Number of Subjects Reported With Unsolicited Adverse Events (AEs)
Description: The outcome measure was not reporting statistics for all the arms in the baseline period. Results were tabulated on baseline groups except for the Synforix PRE and Synforix POST groups, for which results were presented for the Pooled Synforix PRE and POST Group.
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Days 0-30) after primary vaccine dose.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Synflorix PRE and POST Group: Pooled group with subjects from both, Synflorix PRE Group and Synflorix POST Group, that received in this study (before and after the implementation of the protocol amendment) a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa without prophylactic antipyretic treatment.
Arm/Group | Synflorix I Group | Synflorix II Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix PRE and POST Group
Number analyzed (Participants) | 178 | 27 | 336 | 209
Participants | 22 | 3 | 64 | 30

6. Secondary Outcome: Number of Subjects Reported With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the entire study period (Month 0-Month 12)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 178 | 27 | 172 | 37 | 336
Participants | 13 | 5 | 13 | 4 | 30

7. Secondary Outcome: Number of Subjects Reported With AEs Resulting in Rash, New Onset of Chronic Illness (NOCI), Emergency Room (ER) Visits and Non-routine Physician Office Visits.
Description: Results were tabulated only on Mencevax + Infanrix Hexa Group, according to the outcome measure specification of the protocol.
Time Frame: Up to 6 months after vaccination with Mencevax™
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 336
Participants
  Subject(s) with any rash(es) | 7
  Subject(s) with any NOCI(s) | 1
  Subject(s) with any ER visit(s) | 0
  Subject(s) with any visit(s) at physician office | 53

8. Secondary Outcome: Number of Subjects With Antibody Concentrations Against Certain Pneumococcal Serotypes ≥ the Cut Off
Description: Certain pneumococcal serotypes includes pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F). Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations were measured by 22F-inhibition Enzyme-Linked ImmunoSorbent Assay (ELISA).
  The seroprotection cut-off for the assay was ≥ 0.2 microgram per milliliter (μg/mL).
Time Frame: Prior to booster vaccination (PRE), 1 month (M1) and 12 months (M12) post-booster vaccination
Population: The analysis were performed on the According-To-Protocol (ATP) cohort for persistence, which included all subjects of the pneumococcal conjugate primed groups for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 141 | 25 | 168 | 37 | 289
Participants
  ANTI-1 PRE: number analyzed (Participants) | 132 | 25 | 163 | 37 | 284
  ANTI-1 PRE | 74 | 14 | 115 | 27 | 6
  ANTI-1 M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 244
  ANTI-1 M1 | 140 | 24 | 167 | 36 | 5
  ANTI-1 M12: number analyzed (Participants) | 138 | 25 | 167 | 36 | 263
  ANTI-1 M12 | 89 | 11 | 122 | 30 | 11
  ANTI-4 PRE: number analyzed (Participants) | 139 | 25 | 160 | 35 | 289
  ANTI-4 PRE | 123 | 15 | 147 | 31 | 6
  ANTI-4 M1: number analyzed (Participants) | 141 | 24 | 167 | 37 | 261
  ANTI-4 M1 | 141 | 24 | 167 | 37 | 6
  ANTI-4 M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 288
  ANTI-4 M12 | 103 | 14 | 147 | 27 | 20
  ANTI-5 PRE: number analyzed (Participants) | 131 | 25 | 156 | 37 | 277
  ANTI-5 PRE | 102 | 15 | 142 | 30 | 6
  ANTI-5 M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 256
  ANTI-5 M1 | 140 | 23 | 167 | 36 | 10
  ANTI-5 M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 281
  ANTI-5 M12 | 113 | 18 | 159 | 30 | 31
  ANTI-6B PRE: number analyzed (Participants) | 139 | 25 | 164 | 37 | 282
  ANTI-6B PRE | 110 | 13 | 143 | 32 | 1
  ANTI-6B M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 282
  ANTI-6B M1 | 134 | 21 | 166 | 35 | 1
  ANTI-6B M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 289
  ANTI-6B M12 | 97 | 18 | 148 | 30 | 21
  ANTI-7F PRE: number analyzed (Participants) | 136 | 24 | 159 | 35 | 281
  ANTI-7F PRE | 130 | 21 | 156 | 34 | 5
  ANTI-7F M1: number analyzed (Participants) | 140 | 25 | 167 | 37 | 265
  ANTI-7F M1 | 140 | 25 | 167 | 37 | 9
  ANTI-7F M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 283
  ANTI-7F M12 | 132 | 21 | 165 | 36 | 20
  ANTI-9V PRE: number analyzed (Participants) | 127 | 24 | 154 | 35 | 279
  ANTI-9V PRE | 117 | 20 | 152 | 34 | 5
  ANTI-9V M1: number analyzed (Participants) | 141 | 25 | 167 | 37 | 266
  ANTI-9V M1 | 141 | 24 | 167 | 37 | 10
  ANTI-9V M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 285
  ANTI-9V M12 | 129 | 20 | 166 | 35 | 30
  ANTI-14 PRE: number analyzed (Participants) | 136 | 25 | 164 | 37 | 274
  ANTI-14 PRE | 131 | 22 | 159 | 35 | 25
  ANTI-14 M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 261
  ANTI-14 M1 | 140 | 24 | 166 | 36 | 29
  ANTI-14 M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 277
  ANTI-14 M12 | 131 | 21 | 166 | 34 | 63
  ANTI-18C PRE: number analyzed (Participants) | 135 | 25 | 163 | 35 | 275
  ANTI-18C PRE | 118 | 14 | 154 | 29 | 8
  ANTI-18C M1: number analyzed (Participants) | 141 | 25 | 167 | 37 | 269
  ANTI-18C M1 | 141 | 25 | 167 | 37 | 9
  ANTI-18C M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 281
  ANTI-18C M12 | 113 | 18 | 157 | 35 | 29
  ANTI-19F PRE: number analyzed (Participants) | 137 | 25 | 165 | 37 | 278
  ANTI-19F PRE | 128 | 21 | 163 | 36 | 17
  ANTI-19F M1: number analyzed (Participants) | 141 | 25 | 167 | 37 | 269
  ANTI-19F M1 | 138 | 25 | 165 | 37 | 24
  ANTI-19F M12: number analyzed (Participants) | 138 | 25 | 168 | 36 | 283
  ANTI-19F M12 | 135 | 22 | 165 | 36 | 90
  ANTI-23F PRE: number analyzed (Participants) | 136 | 25 | 155 | 35 | 275
  ANTI-23F PRE | 103 | 14 | 132 | 30 | 2
  ANTI-23F M1: number analyzed (Participants) | 140 | 24 | 167 | 37 | 259
  ANTI-23F M1 | 135 | 21 | 163 | 36 | 4
  ANTI-23F M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 289
  ANTI-23F M12 | 115 | 16 | 154 | 33 | 24

9. Secondary Outcome: Antibody Concentrations Against Certain Pneumococcal Serotypes ≥ the Cut Off.
Description: Certain pneumococcal serotypes included pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F).
  Anti-1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F antibody concentrations were measured by 22F-inhibition Enzyme-Linked ImmunoSorbent Assay (ELISA).
  Seropositivity cut-off for the assay was ≥ 0.05 microgram per milliliter (μg/mL).
Time Frame: Prior to booster vaccination (PRE), 1 month (M1) and 12 months (M12) post-booster vaccination
Population: The analysis were performed on the ATP cohort for persistence, which included all subjects of the pneumococcal conjugate primed groups for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 141 | 25 | 168 | 37 | 289
μg/mL
  ANTI-1 PRE: number analyzed (Participants) | 132 | 25 | 163 | 37 | 284
  ANTI-1 PRE | 0.22 [0.19 to 0.25] | 0.18 [0.12 to 0.27] | 0.31 [0.27 to 0.35] | 0.26 [0.19 to 0.35] | 0.03 [0.03 to 0.03]
  ANTI-1 M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 244
  ANTI-1 M1 | 1.67 [1.47 to 1.9] | 1.64 [1.08 to 2.47] | 2.62 [2.3 to 2.99] | 2.97 [2.21 to 3.99] | 0.03 [0.03 to 0.03]
  ANTI-1 M12: number analyzed (Participants) | 138 | 25 | 167 | 36 | 263
  ANTI-1 M12 | 0.26 [0.22 to 0.31] | 0.18 [0.12 to 0.29] | 0.39 [0.34 to 0.45] | 0.41 [0.31 to 0.56] | 0.04 [0.04 to 0.04]
  ANTI-4 PRE: number analyzed (Participants) | 139 | 25 | 160 | 35 | 289
  ANTI-4 PRE | 0.4 [0.35 to 0.45] | 0.24 [0.17 to 0.35] | 0.6 [0.52 to 0.69] | 0.45 [0.35 to 0.58] | 0.03 [0.03 to 0.03]
  ANTI-4 M1: number analyzed (Participants) | 141 | 24 | 167 | 37 | 261
  ANTI-4 M1 | 3.01 [2.69 to 3.36] | 2.84 [1.98 to 4.08] | 4.21 [3.72 to 4.76] | 3.95 [2.97 to 5.26] | 0.03 [0.03 to 0.03]
  ANTI-4 M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 288
  ANTI-4 M12 | 0.34 [0.29 to 0.39] | 0.21 [0.13 to 0.33] | 0.5 [0.43 to 0.56] | 0.55 [0.39 to 0.78] | 0.04 [0.03 to 0.04]
  ANTI-5 PRE: number analyzed (Participants) | 131 | 25 | 156 | 37 | 277
  ANTI-5 PRE | 0.36 [0.32 to 0.42] | 0.31 [0.18 to 0.52] | 0.59 [0.52 to 0.68] | 0.53 [0.36 to 0.78] | 0.04 [0.03 to 0.04]
  ANTI-5 M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 256
  ANTI-5 M1 | 2.3 [2.04 to 2.6] | 2 [1.31 to 3.06] | 3.68 [3.26 to 4.15] | 3.03 [2.16 to 4.26] | 0.04 [0.03 to 0.04]
  ANTI-5 M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 281
  ANTI-5 M12 | 0.42 [0.36 to 0.48] | 0.35 [0.23 to 0.52] | 0.72 [0.63 to 0.83] | 0.58 [0.42 to 0.81] | 0.06 [0.05 to 0.06]
  ANTI-6B PRE: number analyzed (Participants) | 139 | 25 | 164 | 37 | 282
  ANTI-6B PRE | 0.35 [0.3 to 0.41] | 0.18 [0.1 to 0.32] | 0.55 [0.48 to 0.63] | 0.5 [0.35 to 0.72] | 0.03 [0.03 to 0.03]
  ANTI-6B M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 282
  ANTI-6B M1 | 1.35 [1.12 to 1.61] | 0.89 [0.46 to 1.72] | 2.45 [2.17 to 2.77] | 2.25 [1.51 to 3.33] | 0.03 [0.03 to 0.03]
  ANTI-6B M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 289
  ANTI-6B M12 | 0.4 [0.32 to 0.5] | 0.36 [0.19 to 0.66] | 0.56 [0.47 to 0.68] | 0.54 [0.37 to 0.81] | 0.04 [0.04 to 0.04]
  ANTI-7F PRE: number analyzed (Participants) | 136 | 24 | 159 | 35 | 281
  ANTI-7F PRE | 0.74 [0.65 to 0.84] | 0.55 [0.4 to 0.76] | 1.05 [0.93 to 1.18] | 0.87 [0.66 to 1.13] | 0.03 [0.03 to 0.03]
  ANTI-7F M1: number analyzed (Participants) | 140 | 25 | 167 | 37 | 265
  ANTI-7F M1 | 2.9 [2.59 to 3.25] | 2.37 [1.86 to 3.03] | 4.13 [3.69 to 4.63] | 4.38 [3.35 to 5.72] | 0.03 [0.03 to 0.03]
  ANTI-7F M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 283
  ANTI-7F M12 | 0.68 [0.6 to 0.78] | 0.45 [0.32 to 0.63] | 0.91 [0.82 to 1.02] | 0.96 [0.74 to 1.24] | 0.04 [0.04 to 0.04]
  ANTI-9V PRE: number analyzed (Participants) | 127 | 24 | 154 | 35 | 279
  ANTI-9V PRE | 0.61 [0.53 to 0.7] | 0.59 [0.33 to 1.05] | 1 [0.88 to 1.13] | 0.99 [0.78 to 1.26] | 0.03 [0.03 to 0.03]
  ANTI-9V M1: number analyzed (Participants) | 141 | 25 | 167 | 37 | 266
  ANTI-9V M1 | 2.86 [2.52 to 3.23] | 2.57 [1.73 to 3.81] | 4.39 [3.91 to 4.94] | 4.35 [3.3 to 5.73] | 0.03 [0.03 to 0.03]
  ANTI-9V M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 285
  ANTI-9V M12 | 0.67 [0.56 to 0.8] | 0.55 [0.33 to 0.92] | 0.97 [0.85 to 1.12] | 0.86 [0.64 to 1.17] | 0.04 [0.04 to 0.05]
  ANTI-14 PRE: number analyzed (Participants) | 136 | 25 | 164 | 37 | 274
  ANTI-14 PRE | 0.82 [0.69 to 0.96] | 0.52 [0.36 to 0.74] | 1.57 [1.32 to 1.86] | 1.27 [0.86 to 1.88] | 0.04 [0.04 to 0.05]
  ANTI-14 M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 261
  ANTI-14 M1 | 4.58 [4.05 to 5.18] | 4.37 [3.01 to 6.33] | 5.95 [5.28 to 6.71] | 5.86 [4.35 to 7.89] | 0.05 [0.04 to 0.05]
  ANTI-14 M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 277
  ANTI-14 M12 | 0.89 [0.73 to 1.09] | 0.94 [0.48 to 1.84] | 1.54 [1.3 to 1.81] | 1.25 [0.9 to 1.76] | 0.11 [0.09 to 0.13]
  ANTI-18C PRE: number analyzed (Participants) | 135 | 25 | 163 | 35 | 275
  ANTI-18C PRE | 0.47 [0.41 to 0.54] | 0.29 [0.2 to 0.43] | 0.78 [0.69 to 0.89] | 0.54 [0.39 to 0.76] | 0.03 [0.03 to 0.03]
  ANTI-18C M1: number analyzed (Participants) | 141 | 25 | 167 | 37 | 269
  ANTI-18C M1 | 4.96 [4.4 to 5.6] | 3.46 [2.35 to 5.09] | 7 [6.28 to 7.79] | 6.13 [4.85 to 7.75] | 0.03 [0.03 to 0.03]
  ANTI-18C M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 281
  ANTI-18C M12 | 0.56 [0.47 to 0.66] | 0.44 [0.27 to 0.72] | 1.05 [0.92 to 1.21] | 0.92 [0.69 to 1.21] | 0.04 [0.04 to 0.05]
  ANTI-19F PRE: number analyzed (Participants) | 137 | 25 | 165 | 37 | 278
  ANTI-19F PRE | 0.98 [0.81 to 1.19] | 0.63 [0.39 to 1.02] | 1.48 [1.27 to 1.73] | 1.4 [1 to 1.97] | 0.03 [0.03 to 0.04]
  ANTI-19F M1: number analyzed (Participants) | 141 | 25 | 167 | 37 | 269
  ANTI-19F M1 | 6 [5.08 to 7.08] | 4.84 [3.47 to 6.77] | 7.55 [6.48 to 8.79] | 8.77 [6.68 to 11.53] | 0.05 [0.04 to 0.05]
  ANTI-19F M12: number analyzed (Participants) | 138 | 25 | 168 | 36 | 283
  ANTI-19F M12 | 1.46 [1.18 to 1.82] | 0.82 [0.56 to 1.2] | 1.8 [1.52 to 2.13] | 2.04 [1.41 to 2.94] | 0.12 [0.1 to 0.14]
  ANTI-23F PRE: number analyzed (Participants) | 136 | 25 | 155 | 35 | 275
  ANTI-23F PRE | 0.38 [0.31 to 0.46] | 0.3 [0.16 to 0.58] | 0.54 [0.45 to 0.64] | 0.45 [0.31 to 0.65] | 0.03 [0.03 to 0.03]
  ANTI-23F M1: number analyzed (Participants) | 140 | 24 | 167 | 37 | 259
  ANTI-23F M1 | 1.99 [1.67 to 2.38] | 1.33 [0.64 to 2.78] | 2.92 [2.5 to 3.4] | 3.86 [2.52 to 5.91] | 0.03 [0.03 to 0.03]
  ANTI-23F M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 289
  ANTI-23F M12 | 0.46 [0.38 to 0.56] | 0.29 [0.16 to 0.52] | 0.8 [0.67 to 0.95] | 0.98 [0.69 to 1.39] | 0.04 [0.03 to 0.04]

10. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8.
Time Frame: Prior to booster vaccination (PRE), 1 month (M1) and 12 months (M12) post-booster vaccination
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 131 | 25 | 161 | 35 | 135
Titers
  OPSONO-1 PRE: number analyzed (Participants) | 125 | 25 | 152 | 31 | 26
  OPSONO-1 PRE | 6.1 [5 to 7.4] | 5.6 [4 to 8] | 8.1 [6.6 to 10] | 6 [4.2 to 8.5] | 4.9 [3.7 to 6.5]
  OPSONO-1 M1: number analyzed (Participants) | 130 | 23 | 156 | 34 | 39
  OPSONO-1 M1 | 144.6 [109.6 to 190.6] | 193.4 [95.8 to 390.8] | 417 [330.6 to 526.2] | 325 [178.8 to 590.7] | 5.1 [4.1 to 6.4]
  OPSONO-1 M12: number analyzed (Participants) | 129 | 21 | 153 | 34 | 126
  OPSONO-1 M12 | 12.8 [10 to 16.5] | 12.5 [6.8 to 23.2] | 23.1 [18.2 to 29.2] | 20.5 [13.1 to 32.3] | 4.7 [4.3 to 5.1]
  OPSONO-4 PRE: number analyzed (Participants) | 121 | 22 | 148 | 31 | 31
  OPSONO-4 PRE | 23.8 [16.5 to 34.2] | 8.8 [5.2 to 14.9] | 44.9 [33.2 to 60.8] | 29.7 [14.3 to 61.6] | 5.9 [3.4 to 10.2]
  OPSONO-4 M1: number analyzed (Participants) | 130 | 22 | 158 | 32 | 23
  OPSONO-4 M1 | 1547.9 [1357.9 to 1764.4] | 971.6 [615.8 to 1532.7] | 2297 [2005.8 to 2630.4] | 1303.2 [918.6 to 1849] | 7.8 [3.6 to 16.8]
  OPSONO-4 M12: number analyzed (Participants) | 125 | 21 | 152 | 33 | 119
  OPSONO-4 M12 | 19.9 [13.9 to 28.6] | 14.9 [6.4 to 34.8] | 51.2 [36.2 to 72.4] | 72.5 [33.7 to 156.1] | 6.8 [5 to 9.3]
  OPSONO-5 PRE: number analyzed (Participants) | 121 | 24 | 146 | 31 | 26
  OPSONO-5 PRE | 8.5 [7 to 10.4] | 10.4 [6.2 to 17.4] | 16.6 [13.2 to 20.9] | 15.1 [8.8 to 25.9] | 4.2 [3.8 to 4.7]
  OPSONO-5 M1: number analyzed (Participants) | 130 | 23 | 156 | 34 | 45
  OPSONO-5 M1 | 134.3 [109.8 to 164.2] | 105 [55.9 to 196.9] | 289.3 [243.5 to 343.7] | 227.7 [130.7 to 396.6] | 4.3 [3.8 to 4.8]
  OPSONO-5 M12: number analyzed (Participants) | 124 | 21 | 154 | 32 | 135
  OPSONO-5 M12 | 10.3 [8.3 to 12.9] | 10.5 [5.9 to 18.7] | 23.7 [18.9 to 29.8] | 15.4 [10.2 to 23.2] | 4 [4 to 4]
  OPSONO-6B PRE: number analyzed (Participants) | 126 | 22 | 154 | 31 | 25
  OPSONO-6B PRE | 32.5 [21.6 to 48.9] | 15.9 [6 to 42.1] | 45.2 [32.9 to 62.2] | 49.7 [23 to 107.3] | 9.9 [3.5 to 27.7]
  OPSONO-6B M1: number analyzed (Participants) | 130 | 22 | 157 | 34 | 29
  OPSONO-6B M1 | 496.7 [351.4 to 702.2] | 148.3 [46.5 to 472.5] | 985.7 [807.1 to 1203.9] | 718.3 [445.7 to 1157.5] | 20.9 [6.6 to 65.9]
  OPSONO-6B M12: number analyzed (Participants) | 123 | 22 | 145 | 31 | 113
  OPSONO-6B M12 | 46.9 [29.6 to 74.2] | 97.7 [27.7 to 345.1] | 53.9 [36.1 to 80.4] | 29.4 [13.2 to 65.2] | 19.1 [12 to 30.5]
  OPSONO-7F PRE: number analyzed (Participants) | 115 | 22 | 148 | 32 | 23
  OPSONO-7F PRE | 413.6 [266.1 to 642.9] | 221.4 [65.7 to 745.9] | 584.7 [426.1 to 802.3] | 258.4 [119.9 to 556.7] | 90 [23.2 to 349.8]
  OPSONO-7F M1: number analyzed (Participants) | 130 | 23 | 158 | 34 | 28
  OPSONO-7F M1 | 4025.8 [3457.3 to 4687.9] | 1749 [1144.2 to 2673.4] | 4674.7 [4102.2 to 5327] | 2212.2 [1569.1 to 3118.7] | 267.3 [89.1 to 801.2]
  OPSONO-7F M12: number analyzed (Participants) | 130 | 25 | 159 | 34 | 118
  OPSONO-7F M12 | 1503.3 [1209.1 to 1869.2] | 1606.4 [1101.4 to 2343] | 1285.7 [1050.8 to 1573] | 1738.3 [1330.6 to 2271] | 681.1 [499.7 to 928.3]
  OPSONO-9V PRE: number analyzed (Participants) | 119 | 21 | 147 | 31 | 23
  OPSONO-9V PRE | 420.7 [342.7 to 516.5] | 472.9 [255.6 to 874.7] | 407.7 [340.3 to 488.4] | 365.7 [240.6 to 555.8] | 69.2 [22.9 to 208.9]
  OPSONO-9V M1: number analyzed (Participants) | 129 | 23 | 157 | 34 | 31
  OPSONO-9V M1 | 2234.8 [1905.7 to 2620.7] | 752.9 [476.9 to 1188.8] | 2403.7 [2092.3 to 2761.4] | 1155.5 [733.4 to 1820.4] | 87.4 [45.2 to 169]
  OPSONO-9V M12: number analyzed (Participants) | 131 | 25 | 161 | 35 | 124
  OPSONO-9V M12 | 791.6 [647.4 to 967.9] | 552.2 [337.1 to 904.6] | 906.7 [757.6 to 1085.2] | 716.8 [481 to 1068.2] | 127.2 [86.8 to 186.2]
  OPSONO-14 PRE: number analyzed (Participants) | 118 | 21 | 152 | 29 | 12
  OPSONO-14 PRE | 189.7 [141.7 to 254] | 150.2 [81.5 to 276.8] | 293.2 [235.3 to 365.5] | 227.4 [115.1 to 449.4] | 11.5 [3.3 to 40.1]
  OPSONO-14 M1: number analyzed (Participants) | 130 | 22 | 154 | 34 | 19
  OPSONO-14 M1 | 1581.7 [1381.1 to 1811.4] | 1515 [911.2 to 2519] | 1865.2 [1633.4 to 2129.9] | 1964.5 [1359.9 to 2837.9] | 158 [59.4 to 420.2]
  OPSONO-14 M12: number analyzed (Participants) | 117 | 15 | 147 | 32 | 98
  OPSONO-14 M12 | 434.5 [353 to 534.8] | 438.4 [137.7 to 1396] | 447.5 [376 to 532.6] | 558 [425 to 732.5] | 287.8 [203.2 to 407.6]
  OPSONO-18C PRE: number analyzed (Participants) | 124 | 23 | 148 | 24 | 38
  OPSONO-18C PRE | 6.1 [5.2 to 7.2] | 6 [3.7 to 9.7] | 11.7 [9.2 to 15.1] | 9.5 [4.9 to 18.5] | 4.5 [3.5 to 5.8]
  OPSONO-18C M1: number analyzed (Participants) | 128 | 22 | 154 | 34 | 42
  OPSONO-18C M1 | 652.9 [553.5 to 770.1] | 269.7 [128.9 to 564.3] | 737.8 [633.6 to 859.1] | 537.6 [370.9 to 779.3] | 4 [4 to 4]
  OPSONO-18C M12: number analyzed (Participants) | 121 | 23 | 154 | 28 | 124
  OPSONO-18C M12 | 11.9 [8.9 to 16.1] | 24.7 [9 to 67.5] | 27.7 [21.3 to 36] | 23.5 [11 to 50.3] | 4.6 [4 to 5.3]
  OPSONO-19F PRE: number analyzed (Participants) | 121 | 24 | 149 | 32 | 39
  OPSONO-19F PRE | 21.2 [16.1 to 28] | 17.4 [10.5 to 28.7] | 35.1 [28 to 44] | 36.4 [22 to 60.3] | 5.3 [3.7 to 7.7]
  OPSONO-19F M1: number analyzed (Participants) | 130 | 23 | 156 | 34 | 42
  OPSONO-19F M1 | 629.4 [496.6 to 797.7] | 372.9 [180.1 to 772.5] | 1062.2 [871.8 to 1294.3] | 1198.8 [807.1 to 1780.5] | 4.5 [3.7 to 5.6]
  OPSONO-19F M12: number analyzed (Participants) | 130 | 25 | 155 | 35 | 132
  OPSONO-19F M12 | 64.3 [47.6 to 86.7] | 39.4 [17.3 to 89.5] | 101.3 [80.7 to 127] | 121.3 [67.5 to 218.1] | 6.4 [5.1 to 8.1]
  OPSONO-23F PRE: number analyzed (Participants) | 122 | 20 | 149 | 31 | 25
  OPSONO-23F PRE | 288.7 [192.1 to 434] | 310.1 [85.9 to 1119.4] | 408 [288.6 to 576.6] | 305.3 [135 to 690.5] | 20.2 [7.2 to 56.2]
  OPSONO-23F M1: number analyzed (Participants) | 130 | 23 | 157 | 34 | 28
  OPSONO-23F M1 | 2335.7 [2016.2 to 2705.7] | 1223.1 [910.6 to 1642.8] | 3154 [2658 to 3742.4] | 1808.7 [1381.1 to 2368.7] | 261.8 [97.9 to 700.5]
  OPSONO-23F M12: number analyzed (Participants) | 122 | 20 | 152 | 33 | 124
  OPSONO-23F M12 | 386.4 [250 to 597.2] | 433.8 [110.1 to 1709.8] | 857.5 [634 to 1159.7] | 670.2 [331.9 to 1353.3] | 147.1 [86.7 to 249.9]

11. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: The seropositivity cut-off for the assay was ≥ 100 Enzyme-Linked ImmunoSorbent Assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: Prior to booster vaccination (PRE), 1 month (M1) and 12 months (M12) post-booster vaccination
Population: The analyses were performed on the ATP cohort for persistence, which included all subjects of the pneumococcal conjugate primed groups for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 140 | 25 | 167 | 37 | 270
EL.U/mL
  Anti-PD-PRE: number analyzed (Participants) | 135 | 25 | 158 | 37 | 260
  Anti-PD-PRE | 365.1 [302.1 to 441.1] | 356.5 [247 to 514.4] | 685.5 [585.4 to 802.9] | 584.3 [393.1 to 868.4] | 65.6 [60.9 to 70.8]
  Anti-PD-M1: number analyzed (Participants) | 140 | 24 | 166 | 36 | 258
  Anti-PD-M1 | 1654 [1399.9 to 1954.4] | 1813.5 [1111.5 to 2958.9] | 3134.2 [2765.4 to 3552.1] | 2612.3 [1804.4 to 3782.1] | 64.6 [59.9 to 69.5]
  Anti-PD-M12: number analyzed (Participants) | 138 | 25 | 167 | 36 | 270
  Anti-PD-M12 | 468.1 [381.8 to 573.8] | 418 [259.9 to 672.3] | 834.6 [720 to 967.5] | 713.4 [476.9 to 1067.4] | 74.4 [67.8 to 81.6]

12. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes 6A and 19A (Anti-6A and 19A)
Description: Anti-6A and 19A antibody concentrations were measured by 22F-inhibition Enzyme-Linked ImmunoSorbent Assay (ELISA).
Time Frame: Prior to booster vaccination (PRE), 1 month (M1) and 12 months (M12) post-booster vaccination
Population: as for outcome 9
Measure: Geometric Mean (97.5% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 139 | 25 | 168 | 37 | 288
μg/mL
  Anti-6A-PRE: number analyzed (Participants) | 136 | 25 | 161 | 37 | 278
  Anti-6A-PRE | 0.12 [0.1 to 0.15] | 0.08 [0.05 to 0.12] | 0.21 [0.18 to 0.26] | 0.19 [0.12 to 0.29] | 0.03 [0.03 to 0.03]
  Anti-6A-M1: number analyzed (Participants) | 138 | 25 | 166 | 36 | 288
  Anti-6A-M1 | 0.4 [0.31 to 0.51] | 0.29 [0.15 to 0.55] | 0.86 [0.69 to 1.07] | 0.75 [0.43 to 1.3] | 0.03 [0.03 to 0.03]
  Anti-6A-M12: number analyzed (Participants) | 139 | 25 | 167 | 36 | 279
  Anti-6A-M12 | 0.14 [0.11 to 0.18] | 0.1 [0.07 to 0.16] | 0.24 [0.2 to 0.3] | 0.2 [0.13 to 0.29] | 0.04 [0.03 to 0.04]
  Anti-19A-PRE: number analyzed (Participants) | 138 | 25 | 165 | 35 | 277
  Anti-19A-PRE | 0.15 [0.13 to 0.18] | 0.12 [0.07 to 0.19] | 0.23 [0.19 to 0.27] | 0.2 [0.14 to 0.29] | 0.03 [0.03 to 0.04]
  Anti-19A-M1: number analyzed (Participants) | 138 | 25 | 166 | 37 | 276
  Anti-19A-M1 | 0.84 [0.67 to 1.05] | 0.56 [0.29 to 1.09] | 1.34 [1.09 to 1.66] | 1.54 [0.98 to 2.43] | 0.04 [0.03 to 0.04]
  Anti-19A-M12: number analyzed (Participants) | 139 | 25 | 168 | 36 | 284
  Anti-19A-M12 | 0.22 [0.17 to 0.28] | 0.13 [0.08 to 0.22] | 0.36 [0.3 to 0.44] | 0.41 [0.26 to 0.65] | 0.06 [0.05 to 0.07]

13. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: OPA titers against pneumococcal serotypes 6A and 19A (Opsono-6A and 19A) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8.
Time Frame: Prior to booster vaccination (PRE), 1 month (M1) and 12 months (M12) post-booster vaccination
Population: as for outcome 9
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 129 | 22 | 153 | 33 | 131
Titers
  OPSONO-6A-PRE: number analyzed (Participants) | 116 | 19 | 139 | 20 | 24
  OPSONO-6A-PRE | 72.4 [48.3 to 108.4] | 35.6 [12.2 to 104.1] | 65.4 [45.7 to 93.7] | 66 [25.7 to 169.5] | 9.7 [4.7 to 20]
  OPSONO-6A-M1: number analyzed (Participants) | 124 | 21 | 149 | 31 | 16
  OPSONO-6A-M1 | 251.5 [180.2 to 351] | 105.1 [40.6 to 271.8] | 401.7 [319.5 to 505.2] | 403.7 [253.5 to 642.9] | 16.1 [5 to 52]
  OPSONO-6A-M12: number analyzed (Participants) | 111 | 17 | 131 | 29 | 115
  OPSONO-6A-M12 | 59.4 [38.8 to 91] | 23 [8.4 to 62.6] | 52.1 [35.6 to 76.3] | 37.2 [17.5 to 79] | 17.1 [11.7 to 24.9]
  OPSONO-19A-PRE: number analyzed (Participants) | 118 | 21 | 141 | 28 | 36
  OPSONO-19A-PRE | 5 [4.3 to 5.7] | 4.9 [3.2 to 7.3] | 4.8 [4.3 to 5.4] | 5 [3.6 to 6.9] | 4 [4 to 4]
  OPSONO-19A-M1: number analyzed (Participants) | 129 | 18 | 151 | 31 | 45
  OPSONO-19A-M1 | 39.2 [26.4 to 58.2] | 39.7 [11.5 to 137.4] | 89.7 [61.2 to 131.6] | 99.6 [40.8 to 243.1] | 4 [4 to 4]
  OPSONO-19A-M12: number analyzed (Participants) | 127 | 22 | 153 | 33 | 131
  OPSONO-19A-M12 | 7 [5.5 to 8.8] | 4.8 [3.6 to 6.5] | 8.9 [7.1 to 11.1] | 9.5 [5.6 to 16.1] | 4.7 [4.2 to 5.2]

14. Secondary Outcome: Number of Subjects With Serum Bactericidal Antibodies, Using Baby Rabbit Complement for Assay (rSBA) Titres ≥ the Cut-off Values
Description: The cut-off values assessed were 1:8 and 1:128 for meningococcal polysaccharides A , C, W-135 and Y serum bactericidal antibodies, using baby rabbit complement for assay (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY).
  Results were only tabulated for subjects who received a vaccine including the respective antigens (Mencevax + Infanrix Hexa Group).
Time Frame: Prior to vaccination (PRE), 1 month (M1) and 12 months (M12) post-vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all subjects of the pneumococcal conjugate primed groups for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 301
Participants
  rSBA-MenA,Pre, ≥ 1:8: number analyzed (Participants) | 244
  rSBA-MenA,Pre, ≥ 1:8 | 69
  rSBA-MenA, Pre, ≥ 1:128: number analyzed (Participants) | 244
  rSBA-MenA, Pre, ≥ 1:128 | 44
  rSBA-MenA, M1, ≥ 1:8: number analyzed (Participants) | 299
  rSBA-MenA, M1, ≥ 1:8 | 298
  rSBA-MenA, M1, ≥ 1:128: number analyzed (Participants) | 299
  rSBA-MenA, M1, ≥ 1:128 | 298
  rSBA-MenA, M12, ≥ 1:8: number analyzed (Participants) | 136
  rSBA-MenA, M12, ≥ 1:8 | 136
  rSBA-MenA, M12, ≥ 1:128: number analyzed (Participants) | 136
  rSBA-MenA, M12, ≥ 1:128 | 134
  rSBA-MenC,Pre, ≥ 1:8: number analyzed (Participants) | 295
  rSBA-MenC,Pre, ≥ 1:8 | 50
  rSBA-MenC, Pre, ≥ 1:128: number analyzed (Participants) | 295
  rSBA-MenC, Pre, ≥ 1:128 | 17
  rSBA-MenC, M1, ≥ 1:8 | 300
  rSBA-MenC, M1, ≥ 1:128 | 294
  rSBA-MenC, M12, ≥ 1:8: number analyzed (Participants) | 161
  rSBA-MenC, M12, ≥ 1:8 | 154
  rSBA-MenC, M12, ≥ 1:128: number analyzed (Participants) | 161
  rSBA-MenC, M12, ≥ 1:128 | 105
  rSBA-MenW-135,Pre, ≥ 1:8: number analyzed (Participants) | 287
  rSBA-MenW-135,Pre, ≥ 1:8 | 114
  rSBA-MenW-135, Pre, ≥ 1:128: number analyzed (Participants) | 287
  rSBA-MenW-135, Pre, ≥ 1:128 | 59
  rSBA-MenW-135, M1, ≥ 1:8 | 301
  rSBA-MenW-135, M1, ≥ 1:128 | 301
  rSBA-MenW-135, M12, ≥ 1:8: number analyzed (Participants) | 139
  rSBA-MenW-135, M12, ≥ 1:8 | 138
  rSBA-MenW-135, M12, ≥ 1:128: number analyzed (Participants) | 139
  rSBA-MenW-135, M12, ≥ 1:128 | 129
  rSBA-MenY,Pre, ≥ 1:8: number analyzed (Participants) | 297
  rSBA-MenY,Pre, ≥ 1:8 | 167
  rSBA-MenY, Pre, ≥ 1:128: number analyzed (Participants) | 297
  rSBA-MenY, Pre, ≥ 1:128 | 93
  rSBA-MenY, M1, ≥ 1:8 | 300
  rSBA-MenY, M1, ≥ 1:128 | 300
  rSBA-MenY, M12, ≥ 1:8: number analyzed (Participants) | 138
  rSBA-MenY, M12, ≥ 1:8 | 137
  rSBA-MenY, M12, ≥ 1:128: number analyzed (Participants) | 138
  rSBA-MenY, M12, ≥ 1:128 | 127

15. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers in the Mencevax + Infanrix Hexa Group
Description: Results were only tabulated for subjects who received a vaccine including the respective antigens (Mencevax + Infanrix Hexa Group).
Time Frame: Prior to vaccination(PRE), 1 month (M1) and 12 months (M12) post- vaccination.
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 301
Titers
  rSBA-MenA,Pre: number analyzed (Participants) | 244
  rSBA-MenA,Pre | 11.5 [9.2 to 14.3]
  rSBA-MenA, M1: number analyzed (Participants) | 299
  rSBA-MenA, M1 | 2151.3 [1927.4 to 2401.2]
  rSBA-MenA, M12: number analyzed (Participants) | 136
  rSBA-MenA, M12 | 677.6 [579.9 to 791.8]
  rSBA-MenC,Pre: number analyzed (Participants) | 295
  rSBA-MenC,Pre | 6.9 [6 to 8]
  rSBA-MenC, M1 | 811.2 [728 to 904]
  rSBA-MenC, M12: number analyzed (Participants) | 161
  rSBA-MenC, M12 | 191.1 [153.5 to 238]
  rSBA-MenW-135,Pre: number analyzed (Participants) | 287
  rSBA-MenW-135,Pre | 16.3 [13.2 to 20.1]
  rSBA-MenW-135, M1 | 5393.6 [4888.2 to 5951.1]
  rSBA-MenW-135, M12: number analyzed (Participants) | 139
  rSBA-MenW-135, M12 | 573.1 [479.3 to 685.3]
  rSBA-MenY,Pre: number analyzed (Participants) | 297
  rSBA-MenY,Pre | 30.2 [24.2 to 37.7]
  rSBA-MenY, M1 | 2863.7 [2537.8 to 3231.4]
  rSBA-MenY, M12: number analyzed (Participants) | 138
  rSBA-MenY, M12 | 665.2 [547.9 to 807.7]

16. Secondary Outcome: Number of Subjects With Anti-polysaccharide N (Anti-PS) Concentrations ≥ the Cut-off Values
Description: Anti-PS assessed were anti-PS meningitidis serogroup A (anti-PSA), C (anti-PSC), W (anti-PSW-135) and Y (anti-PSY). The cut-offs for anti-PS concentrations were 0.3 μg/mL and 2.0 μg/mL, tabulated for subjects who received a vaccine including the respective antigens (Mencevax + Infanrix Hexa Group).
Time Frame: Prior to vaccination(PRE), 1 month (M1) and 12 months (M12) post-vaccination
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all subjects of the pneumococcal conjugate primed groups for whom assay results were available for antibodies against at least 1 study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 278
Participants
  ANTI-PSA PRE ≥ 0.3 μg/mL: number analyzed (Participants) | 246
  ANTI-PSA PRE ≥ 0.3 μg/mL | 12
  ANTI-PSA PRE ≥ 2.0 μg/mL: number analyzed (Participants) | 246
  ANTI-PSA PRE ≥ 2.0 μg/mL | 1
  ANTI-PSA M1≥ 0.3 μg/mL: number analyzed (Participants) | 272
  ANTI-PSA M1≥ 0.3 μg/mL | 271
  ANTI-PSA M1 ≥ 2.0 μg/mL: number analyzed (Participants) | 272
  ANTI-PSA M1 ≥ 2.0 μg/mL | 271
  ANTI-PSA M12 ≥ 0.3 μg/mL: number analyzed (Participants) | 153
  ANTI-PSA M12 ≥ 0.3 μg/mL | 133
  ANTI-PSA M12 ≥ 2.0 μg/mL: number analyzed (Participants) | 153
  ANTI-PSA M12 ≥ 2.0 μg/mL | 47
  ANTI-PSC PRE ≥ 0.3 μg/mL: number analyzed (Participants) | 269
  ANTI-PSC PRE ≥ 0.3 μg/mL | 3
  ANTI-PSC PRE ≥ 2.0 μg/mL: number analyzed (Participants) | 269
  ANTI-PSC PRE ≥ 2.0 μg/mL | 0
  ANTI-PSC M1 ≥ 0.3 μg/mL | 278
  ANTI-PSC M1≥ 2.0 μg/mL | 277
  ANTI-PSC M12 ≥ 0.3 μg/mL: number analyzed (Participants) | 157
  ANTI-PSC M12 ≥ 0.3 μg/mL | 94
  ANTI-PSC M12 ≥ 2.0 μg/mL: number analyzed (Participants) | 157
  ANTI-PSC M12 ≥ 2.0 μg/mL | 9
  ANTI-PSW-135 PRE ≥ 0.3 μg/mL: number analyzed (Participants) | 236
  ANTI-PSW-135 PRE ≥ 0.3 μg/mL | 1
  ANTI-PSW-135 PRE ≥ 2.0 μg/mL: number analyzed (Participants) | 236
  ANTI-PSW-135 PRE ≥ 2.0 μg/mL | 0
  ANTI-PSW-135 M1 ≥ 0.3 μg/mL: number analyzed (Participants) | 259
  ANTI-PSW-135 M1 ≥ 0.3 μg/mL | 258
  ANTI-PSW-135 M1 ≥ 2.0 μg/mL: number analyzed (Participants) | 259
  ANTI-PSW-135 M1 ≥ 2.0 μg/mL | 234
  ANTI-PSW-135 M12 ≥ 0.3 μg/mL: number analyzed (Participants) | 132
  ANTI-PSW-135 M12 ≥ 0.3 μg/mL | 117
  ANTI-PSW-135 M12 ≥ 2.0 μg/mL: number analyzed (Participants) | 132
  ANTI-PSW-135 M12 ≥ 2.0 μg/mL | 45
  ANTI-PSY PRE ≥ 0.3 μg/mL: number analyzed (Participants) | 261
  ANTI-PSY PRE ≥ 0.3 μg/mL | 3
  ANTI-PSY PRE ≥ 2.0 μg/mL: number analyzed (Participants) | 261
  ANTI-PSY PRE ≥ 2.0 μg/mL | 0
  ANTI-PSY M1 ≥ 0.3 μg/mL: number analyzed (Participants) | 263
  ANTI-PSY M1 ≥ 0.3 μg/mL | 261
  ANTI-PSY M1 ≥ 2.0 μg/mL: number analyzed (Participants) | 263
  ANTI-PSY M1 ≥ 2.0 μg/mL | 249
  ANTI-PSY M12 ≥ 0.3 μg/mL: number analyzed (Participants) | 135
  ANTI-PSY M12 ≥ 0.3 μg/mL | 131
  ANTI-PSY M12 ≥ 2.0 μg/mL: number analyzed (Participants) | 135
  ANTI-PSY M12 ≥ 2.0 μg/mL | 59

17. Secondary Outcome: Geometric Mean Antibody Concentration (GMCs) for Anti-polysaccharide N (Anti-PS) Antibody Concentrations
Description: Anti-PS assessed were Anti-PSA, anti-PSC, anti-PSW-135 and anti-PSY. Results were only tabulated for subjects who received a vaccine including the respective antigens (Mencevax + Infanrix Hexa Group).
Time Frame: Prior to vaccination(PRE), 1 month (M1) and 12 months (M12) post- vaccination.
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 278
μg/mL
  Anti-PSA, Pre: number analyzed (Participants) | 246
  Anti-PSA, Pre | 0.16 [0.15 to 0.17]
  Anti-PSA, M1: number analyzed (Participants) | 272
  Anti-PSA, M1 | 36.28 [32.8 to 40.15]
  Anti-PSA, M12: number analyzed (Participants) | 153
  Anti-PSA, M12 | 0.99 [0.82 to 1.19]
  Anti-PSC, Pre: number analyzed (Participants) | 269
  Anti-PSC, Pre | 0.15 [0.15 to 0.16]
  Anti-PSC, M1 | 14.12 [13 to 15.32]
  Anti-PSC, M12: number analyzed (Participants) | 157
  Anti-PSC, M12 | 0.42 [0.36 to 0.49]
  Anti-PSW-135, Pre: number analyzed (Participants) | 236
  Anti-PSW-135, Pre | 0.15 [0.15 to 0.15]
  Anti-PSW-135, M1: number analyzed (Participants) | 259
  Anti-PSW-135, M1 | 6.11 [5.45 to 6.86]
  Anti-PSW-135, M12: number analyzed (Participants) | 132
  Anti-PSW-135, M12 | 1.21 [0.98 to 1.48]
  Anti-PSY, Pre: number analyzed (Participants) | 261
  Anti-PSY, Pre | 0.15 [0.15 to 0.16]
  Anti-PSY, M1: number analyzed (Participants) | 263
  Anti-PSY, M1 | 8.03 [7.17 to 8.99]
  Anti-PSY, M12: number analyzed (Participants) | 135
  Anti-PSY, M12 | 1.81 [1.5 to 2.19]

18. Secondary Outcome: Anti-tetanus Toxoids (Anti-T) Antibody Concentrations in the Mencevax + Infanrix Hexa Group
Description: The seroprotection cut-off for the assay was ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: Prior to vaccination (Pre)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 266
IU/mL | 0.512 [0.456 to 0.575]

19. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations in the Mencevax + Infanrix Hexa Group
Description: The seroprotection cut-off for the assay was ≥ 10 milli international units per milliliter (mIU/mL). Results were only tabulated for subjects who received a vaccine including the respective antigens (Mencevax + Infanrix Hexa Group). Dummy lower limit (LL) (0.0) and upper limit UL (99999.9) were entered when number of subjects analysed = 1.
Time Frame: Prior to vaccination (Pre)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 2
mIU/mL | 1336.1 [52.3 to 34160.2]

20. Secondary Outcome: Concentrations of Antibodies Against Diphtheria and Tetanus Toxoids (Anti-D and T).
Description: The seroprotection cut-off for the assay was ≥ 0.1 international units per milliliter (IU/mL).
Time Frame: 1 month post-vaccination (M1)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 140 | 24 | 167 | 37 | 245
IU/mL
  Anti-D, M1: number analyzed (Participants) | 140 | 24 | 166 | 37 | 245
  Anti-D, M1 | 10.112 [9.042 to 11.309] | 9.839 [7.475 to 12.95] | 12.285 [11.18 to 13.5] | 11 [8.786 to 13.77] | 7.291 [6.592 to 8.064]
  Anti-T, M1: number analyzed (Participants) | 139 | 24 | 167 | 37 | 245
  Anti-T, M1 | 7.382 [6.639 to 8.208] | 8.684 [6.37 to 11.839] | 9.583 [8.927 to 10.287] | 8.196 [6.829 to 9.837] | 11.79 [10.684 to 13.011]

21. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: The seropositivity cut-off for the assay was ≥ 5 Enzyme-Linked ImmunoSorbent Assay (ELISA) units per millimiter (EL.U/mL).
Time Frame: 1 month post-vaccination (M1)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 140 | 24 | 167 | 37 | 251
EL.U/mL
  Anti-PT, M1: number analyzed (Participants) | 138 | 24 | 166 | 36 | 248
  Anti-PT, M1 | 83.3 [73.8 to 94] | 81.6 [62.2 to 106.9] | 82 [73.4 to 91.7] | 76.7 [62.2 to 94.4] | 163.1 [143 to 185.9]
  Anti-FHA, M1 | 467.9 [422.4 to 518.3] | 431.1 [318.8 to 582.9] | 453.8 [412.6 to 499.1] | 400.4 [321.8 to 498.2] | 580.8 [532.2 to 633.8]
  Anti-PRN, M1: number analyzed (Participants) | 140 | 24 | 167 | 36 | 246
  Anti-PRN, M1 | 222.8 [193.9 to 256] | 153.4 [97.5 to 241.2] | 254.9 [225.8 to 287.8] | 220.4 [168.7 to 288] | 350.7 [316.8 to 388.3]

22. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations
Description: The seroprotection cut-off for the assay was ≥ 10 mIU/mL.
Time Frame: 1 month post-vaccination (M1)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 105 | 16 | 130 | 26 | 1
mIU/mL | 1883.9 [1332.9 to 2662.7] | 1460.6 [816.4 to 2613.2] | 2133 [1615 to 2817.1] | 1818.5 [1142.8 to 2893.6] | 20610 [NA to NA] — As there was only 1 subject analyzed, the lower and upper limits were not quantifiable.

23. Secondary Outcome: Anti-polyribosyl-ribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: The seroprotection cut-off for the assay was ≥ 0.15 μg/mL.
Time Frame: 1 month post-vaccination (M1)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- Synflorix I Group: Subjects were vaccinated with 3 primary vaccination doses of 10Pn vaccine with prophylactic administration of paracetamol in study 10PN-PD-DIT-010 (107017), and received in this study at 12-15 months of age a booster dose of Synforix™ vaccine, co-administered with Infanrix™ hexa along with prophylactic antipyretic treatment.
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 141 | 24 | 167 | 36 | 269
μg/mL | 23.066 [18.806 to 28.291] | 26.006 [15.56 to 43.463] | 27.373 [22.915 to 32.697] | 22.011 [16.288 to 29.745] | 20.985 [17.966 to 24.511]

24. Secondary Outcome: Anti-poliovirus (Anti-Polio) Types 1, 2 and 3 Titers
Description: The seroprotection cut-off for the assay was ≥ 8.
Time Frame: 1 month post-vaccination (M1)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 93 | 12 | 114 | 23 | 1
Titers
  Anti-Polio 1, M1 | 1193 [993.8 to 1432.2] | 1534.2 [952 to 2472.5] | 1058.7 [870.2 to 1288] | 1208.6 [764.2 to 1911.2] | 4096 [NA to NA] — As there was only 1 subject analyzed, the lower and upper limits were not quantifiable.
  Anti-Polio 2, M1: number analyzed (Participants) | 93 | 12 | 113 | 23 | 1
  Anti-Polio 2, M1 | 1354.1 [1115.8 to 1643.3] | 2047.9 [1246 to 3365.9] | 1413.2 [1174.3 to 1700.7] | 2215.8 [1544.4 to 3178.9] | 8192 [NA to NA] — As there was only 1 subject analyzed, the lower and upper limits were not quantifiable.
  Anti-Polio 3, M1: number analyzed (Participants) | 92 | 12 | 114 | 23 | 1
  Anti-Polio 3, M1 | 2354.2 [1946.1 to 2847.9] | 2233.3 [1300.9 to 3834] | 2647.5 [2221.5 to 3155.3] | 3576.5 [2617.3 to 4887.2] | 8192 [NA to NA] — As there was only 1 subject analyzed, the lower and upper limits were not quantifiable.

25. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations
Description: The seroprotection cut-off for the assay was ≥ 10 mIU/mL.
Time Frame: 12 month post-vaccination (M12)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 107 | 16 | 133 | 20 | 19
mIU/mL | 219.3 [164.8 to 291.7] | 147.3 [62.6 to 346.9] | 231.2 [179.7 to 297.6] | 139.2 [74.3 to 260.9] | 535.1 [277.8 to 1030.6]

26. Secondary Outcome: Anti-poliovirus (Anti-Polio) Type 1, 2 and 3 Titers
Description: The seroprotection cut-off for the assay was ≥ 8.
Time Frame: 12 month post-vaccination (M12)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 97 | 13 | 122 | 14 | 9
Titers
  Anti-Polio 1, M12 | 208.2 [164.7 to 263.2] | 150.4 [87.2 to 259.3] | 234.5 [189.5 to 290.3] | 220.8 [92.3 to 528.2] | 335.4 [146.4 to 768.2]
  Anti-Polio 2, M12: number analyzed (Participants) | 96 | 13 | 122 | 14 | 9
  Anti-Polio 2, M12 | 311.2 [241.5 to 401] | 212.4 [100.5 to 449] | 310.6 [256 to 376.9] | 400 [218.6 to 732.1] | 322.7 [172.9 to 602.3]
  Anti-Polio 3, M12 | 431.3 [332.4 to 559.5] | 301 [125.8 to 720.4] | 506.3 [406.3 to 630.7] | 672.2 [330 to 1369.4] | 203.3 [63.7 to 649.2]

27. Secondary Outcome: Number of Nasopharyngeal Swabs With S.Pneumoniae (Vaccine Serotypes)
Description: Results were tabulated on Pooled Synflorix Group and on Mencevax + Infanrix Hexa Group.
Time Frame: Prior to vaccination(Pre), 1 month post-vaccination (M1), 3 months post-vaccination (M3), 7 months post-vaccination (M7), 12 months post-vaccination (M12) and across all time points (Overall)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Swabs
Groups:
- Pooled Synflorix Group: For carriage analyses the Synforix I, Synforix II, Synflorix PRE Group and Synflorix POST Group were pooled.
Arm/Group | Pooled Synflorix Group | Mencevax + Infanrix Hexa Group
Number analyzed (Participants) | 414 | 336
Swabs
  Pre: number analyzed (Participants) | 407 | 330
  Pre | 43 | 53
  M1: number analyzed (Participants) | 408 | 332
  M1 | 45 | 47
  M3: number analyzed (Participants) | 408 | 332
  M3 | 49 | 55
  M7: number analyzed (Participants) | 406 | 334
  M7 | 42 | 50
  M12: number analyzed (Participants) | 409 | 334
  M12 | 34 | 43
  Overall | 111 | 115

28. Secondary Outcome: Number of Nasopharyngeal Swabs With S.Pneumoniae (Cross-reactive Serotypes)
Description: Results were tabulated on Pooled Synflorix Group and on Mencevax + Infanrix Hexa Group.
Time Frame: as for outcome 27
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Swabs
Arm/Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix Group
Number analyzed (Participants) | 336 | 414
Swabs
  Pre: number analyzed (Participants) | 330 | 407
  Pre | 13 | 15
  M1: number analyzed (Participants) | 332 | 408
  M1 | 19 | 22
  M3: number analyzed (Participants) | 332 | 408
  M3 | 21 | 27
  M7: number analyzed (Participants) | 334 | 406
  M7 | 19 | 21
  M12: number analyzed (Participants) | 334 | 409
  M12 | 19 | 18
  Overall | 55 | 59

29. Secondary Outcome: Number of Nasopharyngeal Swabs With S.Pneumoniae (Non-vaccine and Non-cross-reactive Serotypes)
Description: Results were tabulated on Mencevax + Infanrix Hexa Group and on Pooled Synflorix Group.
Time Frame: as for outcome 27
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Swabs
Arm/Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix Group
Number analyzed (Participants) | 336 | 414
Swabs
  Pre: number analyzed (Participants) | 330 | 407
  Pre | 26 | 27
  M1: number analyzed (Participants) | 332 | 408
  M1 | 30 | 42
  M3: number analyzed (Participants) | 334 | 406
  M3 | 32 | 45
  M7: number analyzed (Participants) | 334 | 406
  M7 | 29 | 42
  M12: number analyzed (Participants) | 334 | 409
  M12 | 22 | 39
  Overall | 82 | 111

30. Secondary Outcome: Number of Nasopharyngeal Swabs With H. Influenzae
Description: Results were tabulated on Mencevax + Infanrix Hexa Group and on Pooled Synflorix Group.
Time Frame: as for outcome 27
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Swabs
Arm/Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix Group
Number analyzed (Participants) | 336 | 414
Swabs
  Pre: number analyzed (Participants) | 312 | 397
  Pre | 41 | 48
  M1: number analyzed (Participants) | 318 | 402
  M1 | 39 | 56
  M3: number analyzed (Participants) | 328 | 403
  M3 | 34 | 62
  M7: number analyzed (Participants) | 332 | 403
  M7 | 49 | 64
  M12: number analyzed (Participants) | 333 | 406
  M12 | 57 | 46
  Overall | 124 | 160

31. Secondary Outcome: Number of Nasopharyngeal Swabs With S. Pneumoniae and H. Influenzae
Description: Results were tabulated on Mencevax + Infanrix Hexa Group and on Pooled Synflorix Group.
Time Frame: as for outcome 27
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Number; unit: Swabs
Arm/Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix Group
Number analyzed (Participants) | 336 | 414
Swabs
  Pre: number analyzed (Participants) | 312 | 397
  Pre | 19 | 21
  M1: number analyzed (Participants) | 318 | 402
  M1 | 20 | 30
  M3: number analyzed (Participants) | 328 | 403
  M3 | 17 | 31
  M7: number analyzed (Participants) | 332 | 403
  M7 | 22 | 28
  M12: number analyzed (Participants) | 333 | 406
  M12 | 22 | 19
  Overall | 61 | 86

32. Secondary Outcome: Number of Subjects With New Acquisition Associated to S. Pneumoniae Detected in Nasopharyngeal Swabs
Description: Results were tabulated on Mencevax + Infanrix Hexa Group and on Pooled Synflorix Group.
Time Frame: 1 month post-vaccination (M1), 3 months post-vaccination (M3), 7 months post-vaccination (M7), 12 months post-vaccination (M12) and across all time points (Overall)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix Group
Number analyzed (Participants) | 336 | 414
Participants
  M1: number analyzed (Participants) | 332 | 408
  M1 | 43 | 56
  M3: number analyzed (Participants) | 332 | 408
  M3 | 63 | 76
  M7: number analyzed (Participants) | 334 | 406
  M7 | 70 | 73
  M12: number analyzed (Participants) | 334 | 409
  M12 | 65 | 70
  Overall | 161 | 195

33. Secondary Outcome: Number of Subjects With New Acquisition Associated to H. Influentzae Detected in Nasopharyngeal Swabs.
Description: Results were tabulated on Mencevax + Infanrix Hexa Group and on Pooled Synflorix Group.
Time Frame: as for outcome 32
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax + Infanrix Hexa Group | Pooled Synflorix Group
Number analyzed (Participants) | 336 | 414
Participants
  M1: number analyzed (Participants) | 318 | 402
  M1 | 21 | 32
  M3: number analyzed (Participants) | 328 | 403
  M3 | 22 | 40
  M7: number analyzed (Participants) | 332 | 403
  M7 | 37 | 42
  M12: number analyzed (Participants) | 333 | 406
  M12 | 39 | 35
  Overall | 104 | 129

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited symptoms: during the 31-day (Days 0-30) follow-up periods after vaccination; SAEs: during the entire study period (from Month 0 up to Month 12).
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix PRE Group | Synflorix POST Group | Mencevax + Infanrix Hexa Group
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/27 | 0/172 | 0/37 | 0/336
Serious Adverse Events (participants affected / at risk) | 13/178 | 5/27 | 13/172 | 4/37 | 30/336
Other Adverse Events (participants affected / at risk) | 153/178 | 23/27 | 154/172 | 35/37 | 290/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix I Group (N=178) | Synflorix II Group (N=27) | Synflorix PRE Group (N=172) | Synflorix POST Group (N=37) | Mencevax + Infanrix Hexa Group (N=336)
Concussion (Infections and infestations) | 1 | 0 | 2 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Caustic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pharyngeal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Testicular retraction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 1 | 4
Laryngitis (Infections and infestations) | 2 | 1 | 1 | 0 | 4
Bronchopneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 2
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 1 | 3
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix I Group (N=178) | Synflorix II Group (N=27) | Synflorix PRE Group (N=172) | Synflorix POST Group (N=37) | Mencevax + Infanrix Hexa Group (N=336)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 47 (47) | 8 (8) | 46 (46) | 10 (10) | 88 (88)
Erythema (Skin and subcutaneous tissue disorders) | 89 (89) | 9 (9) | 74 (74) | 12 (12) | 146 (146)
Irritability (Psychiatric disorders) | 86 (86) | 17 (17) | 105 (105) | 19 (19) | 147 (147)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 3 (3)
Pain (General disorders) | 54 (54) | 10 (10) | 79 (79) | 19 (19) | 114 (114)
Pyrexia (General disorders) | 64 (64) | 14 (14) | 100 (100) | 16 (16) | 146 (147)
Somnolence (Nervous system disorders) | 91 (91) | 11 (11) | 84 (84) | 18 (18) | 146 (146)
Swelling (General disorders) | 52 (52) | 8 (8) | 50 (50) | 13 (13) | 71 (71)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.